CLINICAL TRIAL: NCT05672017
Title: Sweet Consumption and Subsequent Sweet Food Preferences and Intakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AppletonRSFC2022
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Dietary Behaviour

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, outcome assessors and analysts will be masked. It is not possible to mask participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Instructions: Increase sweet food consumption (Active Comparator): Participants are asked to increase their consumption of sweet foods throughout their diet. Participants will be provided with clear instructions, where sweet foods will be highlighted and additional means of increasing sweet food consumption will be offered.
  Interventions: Behavioral: Dietary Instructions
- Dietary Instructions: Decrease sweet food consumption (Active Comparator): Participants are asked to decrease their consumption of sweet foods throughout their diet. Participants will be provided with clear instructions, where sweet foods will be highlighted and means of decreasing sweet food consumption will be offered.
  Interventions: Behavioral: Dietary Instructions
- Dietary Instructions: Usual Diet (Placebo Comparator): Participants are asked to retain their consumption of sweet foods throughout their diet.
  Interventions: Behavioral: Dietary Instructions

INTERVENTIONS:
Behavioral: Dietary Instructions — Dietary Instructions

SUMMARY:
This study will assess the effects of repeated sweet versus non-sweet food consumption on subsequent sweet and non-sweet food preferences and intakes.

DETAILED DESCRIPTION:
Participants will be randomized to receive instructions to either increase, decrease or make no change to sweet food consumption for 6 days, and impacts on food preferences and intakes will be assessed at baseline and after 1 week. Preferences for sweet and non-sweet foods will be assessed during a taste test at each assessment time, where six different foods will be rated. Sweet and non-sweet food consumption will also be measured at a subsequent breakfast at the assessment time. Buffet meals composed of sweet and non-sweet foods suitable for consumption at breakfast will be provided ad-libitum.

A subset of participants (selected at random) (10 participants randomized to increase sweet food consumption and 10 participants randomized to decrease sweet food consumption) will also be assessed via MRI and fMRI scanning to investigate brain structure and functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 years;
2. habitually consume breakfast;
3. able to provide consent and complete all study materials;
4. able to attend Bournemouth University for testing.

Exclusion criteria:

1. individuals who are pregnant or breastfeeding;
2. underweight (BMI <18.5);
3. have pre-existing clinical conditions such as diabetes mellitus, eating disorders, Crohn's disease and other illness's leading to participants receiving external nutritional advice and dietary restrictions;
4. have pre-existing medical conditions affecting swallow ability, taste and smell perception;
5. currently or within 3 months of starting the study are following a specific dietary programme (e.g.: Slimming World);
6. current smokers or have smoked within 3 months of the study start date.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Appleton, Principal Investigator — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, US and Canada Only, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data will be available on completion of the trial from the PI
Supporting Information: Study Protocol, SAP
Time Frame: On study completion
Access Criteria: On reasonable request

REFERENCES:
- [Background] This project is associated with Clinical Trails Registration: NCT03427658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
Started | 40 | 43 | 21
Completed | 40 | 43 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet | Total
Number analyzed (Participants) | 40 | 43 | 21 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (6.4) | 25.3 (6.7) | 20.6 (1.5) | 23.9 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 16 | 75
  Male | 11 | 13 | 5 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 40 | 43 | 21 | 104

OUTCOME MEASURES:

1. Primary Outcome: Sweet Food Preferences
Description: Preferences for various sweet foods/fluids, assessed using a taste test, where participants sample several sweet and non-sweet foods and rate them for pleasantness on a 100mm Visual Analogue Scale, from 0 to 100mm. Higher scores signify stronger preferences
Time Frame: Week 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
Number analyzed (Participants) | 40 | 43 | 21
score on a scale | 66 (3) | 63 (3) | 68 (3)

2. Primary Outcome: Sweet Food Choices
Description: Selection of sweet foods/fluids at a given meal, assessed where participants can consume freely from a meal composed of sweet and non-sweet foods, and proportion of sweet foods consumed is measured as a percentage of weight consumed
Time Frame: Week 1
Measure: Mean (Standard Error); unit: percentage of weight consumed
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
Number analyzed (Participants) | 40 | 43 | 21
percentage of weight consumed | 36 (4) | 25 (4) | 27 (4)

3. Secondary Outcome: Hunger and Thirst
Description: Ratings of subjective perceptions, assessed using 100mm VAS from 0 (lower hunger) to 100 (higher hunger) mm
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
Number analyzed (Participants) | 40 | 43 | 21
score on a scale | 57 (18) | 65 (20) | 64 (18)

4. Secondary Outcome: Sweet Food Perceptions
Description: Perceptions for various sweet foods/fluids, assessed using a taste test, where participants sample several sweet and non-sweet foods and rate them for intensity on a 100mm Visual Analogue Scale from 0 to 100mm. Higher scores signify stronger perceptions
Time Frame: Week 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
Number analyzed (Participants) | 40 | 43 | 21
score on a scale | 71 (3) | 77 (3) | 73 (3)

5. Secondary Outcome: MRI Static Brain Scan (Subset of Participants Only)
Description: Static brain scan gained from a 3-Tesla Siemens Magnetom Lumina scanner (Siemens Healthcare, Erlangen, Germany), used to investigate brain structure, where the anatomical structure (e.g. size, shape) of the brain, measured via surface area (mm squared), will be compared at baseline and week 1
Time Frame: Baseline to week 1
Reporting Status: Not Posted

6. Secondary Outcome: fMRI Composite Functional Brain Scan (Subset of Participants Only)
Description: Composite fMRI functional scan to investigate brain functionality and connectivity in response to a 10 min cognitive task, will be gained from a 3-Tesla Siemens Magnetom Lumina scanner (Siemens Healthcare, Erlangen, Germany), where patterns of activity will be measured using blood oxygenation level-dependent (BOLD) contrast whole-brain functional images, acquired using a T2-weighted gradient-echo Echo Planar Imaging (EPI) sequence and a 32-channel head coil during a 10 min cognitive task, and will be compared at baseline and week 1 (for full details of this methodology see Yankouskaya A, et al., Biology, 2023, 12, 211.)
Time Frame: Baseline to week 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 week
Description: self-report
Arm/Group | Dietary Instructions: Increase Sweet Food Consumption | Dietary Instructions: Decrease Sweet Food Consumption | Dietary Instructions: Usual Diet
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/21
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05672017/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT05672017/SAP_000.pdf